CLINICAL TRIAL: NCT00121095
Title: Phase I/II Trial of Samarium Sm-153 Lexidronam Combined With Docetaxel for Patients With Androgen-Independent Prostate Cancer
Brief Title: Study of Samarium Sm-153 Lexidronam Combined With Docetaxel for Patients With Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cytogen Corporation (Industry)
Responsible Party: Michael Manyak, MD, Cytogen Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 424Sm32
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — samarium Sm-153 lexidronam; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Samarium Sm-153 lexidronam + Docetaxel

INTERVENTIONS:
Drug: Samarium Sm-153 lexidronam + Docetaxel — 1 mCi/kg Sm153 + 75 mg/m2 docetaxel

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and anti-tumor effects of treatment with samarium Sm-153 lexidronam in combination with docetaxel in patients with castrate metastatic prostate cancer.

DETAILED DESCRIPTION:
The principal objective of this trial is to evaluate the safety, feasibility, and anti-tumor effects of a novel bone-targeted regimen consisting of Samarium Sm-153 lexidronam combined with docetaxel and prednisone. This present study design permits evaluation of the clinical activity of combining two distinct agents that have shown benefit for the treatment of patients with advanced androgen-independent prostate cancer and bone metastases. It enables assessment of potential synergistic interactions between a cytotoxic chemotherapy agent and a bone-targeting radioisotope agent in the setting of a bone-targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have histological evidence of adenocarcinoma of the prostate.
* Have progressive castrate metastatic disease.
* Castrate levels of testosterone (<50 ng/ml). Treatment to maintain castrate levels of testosterone must be continued.
* Must have evidence of at least 3 bone metastases on bone scan.
* Patients for whom initial hormone treatment (exclusive of neoadjuvant hormone therapy) was a combined androgen blockade approach, must show progression of disease following withdrawal of the anti-androgen prior to enrollment.
* Patients undergoing prior bisphosphonate treatments are eligible.
* Patients who have received one prior treatment with 153Sm lexidronam or 89Sr are eligible provided it is at least 12 weeks from treatment with 153Sm lexidronam or 24 weeks from treatment with 89Sr.
* Life expectancy of at least 12 weeks (based on co-morbidity).
* KPS>60.
* Lab requirements:

  * White Blood Count (WBC) ≥ 3,000/mm3;
  * Absolute Neutrophil Count (ANC) ≥ 1,500/ mm3;
  * Platelet (PLT) ≥ 100,000/mm3;
  * Hemoglobin (HGB) ≥ 10 mg/dl;
  * Bilirubin ≤ 2.0 mg/dl;
  * ALT/AST≤ 3 times the upper limit of normal;
  * Serum creatinine ≤ 2.0 mg/dl.
* Patients must sign an informed consent.

Exclusion Criteria:

* Patients with small cell carcinoma.
* Patients with predominant visceral metastases (>3 lung or liver lesions) or symptomatic lymphadenopathy (scrotal or pedal edema).
* Patients who have received more than one course of external beam radiation therapy directed at bone lesions.
* Clinically significant cardiac disease (New York Heart Association Class III/IV).
* History of other malignancies (other than non-melanoma skin cancer), unless in complete remission or off therapy for that disease for at least five years.
* Have or are participating in a research study protocol or clinical trial protocol within 30 days of the date of the baseline visit.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2005-07; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Primary outcome is safety and tolerability of the combination treatment

SECONDARY OUTCOMES:
Tumor response will be assessed when possible using RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Morris, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States